CLINICAL TRIAL: NCT04374071
Title: Early Short Course Corticosteroids in Hospitalized Patients With COVID-19
Brief Title: Early Short Course Corticosteroids in COVID-19
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mayur Ramesh, Senior Staff Physician, Infectious Diseases, Henry Ford Health System
Other Study IDs: HFH IRB # 13739
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID; Pneumonia, Viral
Keywords: methyprednisolone
MeSH Terms: conditions — Pneumonia, Viral | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-Corticosteroid protocol: Patients with moderate or severe disease who presented to HFHS within the first week of the COVID epidemic in Detroit were initially treated with supportive care with or without a combination of lopinavir-ritonavir and ribavirin or hydroxychloroquine according an institutional guideline developed by Infectious Diseases Physicians and Pharmacists. The institutional guidelines were developed by consensus, and based on the available literature, experience from Wuhan, China and other centers around the world affected by COVID-19 before Michigan. Intravenous (IV) remdesivir compassionate use was requested for eligible mechanically ventilated patients. On March 17, 2020 lopinavir-ritonavir with ribavirin was removed from the COVID-19 institutional protocol.
- Corticosteroid Protocol: As a result of observed poor outcomes, clinical rationale based upon immunology, clinical course of COVID-19, and more recently best available evidence, the HFHS corticosteroid protocol was developed. We hypothesized that early corticosteroids would combat the inflammatory cascade leading to respiratory failure, ICU escalation of care, and mechanical ventilation. The corticosteroid protocol became the institutional standard on March 20, 2020. Patients with confirmed influenza infection were not recommended to receive corticosteroids.
  Patients with moderate COVID-19 who required 4 liters or more of oxygen per minute on admission, or who had escalating oxygen requirements from baseline, were recommended to receive IV methylprednisolone 0.5 to 1 mg/kg/day in 2 divided doses for 3 days. Patients who required ICU admission were recommended to receive the above regimen of hydroxychloroquine and IV methylprednisolone 0.5 to 1 mg/kg/day in 2 divided doses for 3 to 7 days.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — IV methylprednisolone 0.5 to 1 mg/kg/day in 2 divided doses for 3 days
  Other Names: Corticosteorids
  Groups: Corticosteroid Protocol

SUMMARY:
The investigators intend to study the role of early use of methylprednisolone in the hospitalized patients with a diagnosis of COVID-19 pneumonia.

DETAILED DESCRIPTION:
Consecutive patients hospitalized between March 12, 2020 through March 27, 2020 are eligible for inclusion if they were 18 years of age or older, had confirmed COVID-19 infection, with radiographic evidence of bilateral pulmonary infiltrates, and required oxygen by nasal cannula, high-flow nasal cannula (HFNC), or mechanical ventilation. Patients are excluded if they were transferred from an out-of-system hospital, died within 24 hours of presentation to the ED, or were admitted for less than 24 hours. A confirmed case of COVID-19 was defined as a patient that had a positive reverse-transcriptase-polymerase- chain-reaction (RT-PCR) assay for SARS-CoV-2 in a nasopharyngeal sample.

Patients are risk stratified by severity of symptoms on presentation to the hospital as mild, moderate, or severe COVID-19. Patients without hypoxia or exertional dyspnea were considered to have mild COVID-19. Patients with mild COVID-19 were treated with symptom relief only and not admitted to the hospital. Patients who presented with infiltrates on chest radiography and required supplemental oxygen by nasal cannula or HFNC were classified as having moderate COVID-19. Patients who had respiratory failure requiring mechanical ventilation were classified as having severe COVID-19.

This is a multi-center quasi-experimental study at HFHS, comprised of five hospitals in southeast and south-central Michigan. The study was approved by the institution's Investigational Review Board (#13739) with waiver of consent. Patients in the pre-corticosteroid protocol group from March 12, 2020 through March 19, 2020 were compared to a corticosteroid protocol group that included patients from March 20, 2020 through March 27, 2020.

Patients in both study groups received standard care, comprised of supplemental oxygen, HFNC, invasive ventilation, antibiotic agents, antiviral agents, vasopressor support, and renal-replacement therapy, as determined by the primary team. Patients who progressed to ARDS were managed with standard of care.

Data was ascertained from each institution's electronic medical record and recorded in a standardized electronic case report form. Demographic data, information on clinical symptoms or signs at presentation, and laboratory and radiologic results during admission. All laboratory tests and radiologic assessments, including plain chest radiography and computed tomography of the chest, were performed at the discretion of the treating physician.

Coexisting conditions were ascertained from electronic medical record and physician documentation. The National Early Warning Score (NEWS) was collected to evaluate baseline illness severity based on vital signs obtained in the Emergency Department. Additionally, the quick Sequential Organ Failure Assessment (qSOFA) was used to evaluate severity of illness of included patients based on ED vitals and examination. All patients were followed for at least 14 days after initial presentation. Patient data was censored on April 9, 2020.

Statistical Analysis: Continuous variables were reported as median and interquartile range (IQR) and compared using the Mann-Whitney test or t-test, as appropriate. Categorical data was reported as number and percentage (no., %) and compared using the chi-squared test or Fisher's exact test, as appropriate. No imputation was made for missing data points. The sample size was derived from all eligible consecutive hospitalized patients during the study period. A two-sided α < 0.05 was considered statistically significant. Bivariate and multivariable logistic regression analysis was planned a-priori to test the association between the composite endpoint and exposure to the corticosteroid protocol. Covariates in the bivariate analysis with a p-value <0.2 and clinical rationale were included in a multivariable regression model that was restricted to a subject-to-variable ratio of 10:1. Statistical analysis was performed using IBM SPSS version 25 (Chicago, IL) and SAS 9.4 (Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed COVID-19 infection
* Radiographic evidence of bilateral pulmonary infiltrates
* Oxygen requirement by nasal cannula, high-flow nasal cannula (HFNC), or mechanical ventilation

Exclusion Criteria:

* Transfer from an out-of-system hospital
* Death within 24 hours of presentation to the ED
* Admitted for less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized with confirmed COVID-19 between March 12, 2020 through March 27, 2020 were eligible for inclusion.
  Risk stratification by severity of symptoms on presentation: Patients without hypoxia or exertional dyspnea were considered to have mild COVID-19 and not admitted to the hospital. Patients who presented with infiltrates on chest radiography and required supplemental oxygen by nasal cannula or HFNC were classified as having moderate COVID-19. Patients who had respiratory failure requiring mechanical ventilation were classified as having severe COVID-19.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Transfer to Intensive care unit (ICU) | 14 days followup for every patient in each group
  Number of patients transferred to ICU is each of the groups
Need for Mechanical Ventilation | 14 days followup for every patient in each group
  Number of patients that needed mechanical ventilation in each of the groups
Mortality | 14 days followup for every patient in each group
  Number of patients who died in each of the groups

SECONDARY OUTCOMES:
Development and Severity of ARDS | 14 days followup for every patient in each group
  Number of patients who developed ARDS of varying severity per Berlin classification in each of the groups
Length of hospital stay (LOS). | 14 days followup for every patient in each group
  LOS in each of the groups

CONTACTS AND LOCATIONS:
Overall Officials: Mayur Ramesh, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared One year from publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: One year from publication
Access Criteria: All requests for IPD should be referred to the PI by email.

REFERENCES:
- [Derived] Fadel R, Morrison AR, Vahia A, Smith ZR, Chaudhry Z, Bhargava P, Miller J, Kenney RM, Alangaden G, Ramesh MS; Henry Ford COVID-19 Management Task Force. Early Short-Course Corticosteroids in Hospitalized Patients With COVID-19. Clin Infect Dis. 2020 Nov 19;71(16):2114-2120. doi: 10.1093/cid/ciaa601. PMID 32427279